CLINICAL TRIAL: NCT02715115
Title: A Randomized, Double-blind, Placebo-controlled, Dose-ranging Study of the Safety and Pharmacokinetics of Oral NNZ-2566 in Pediatric Rett Syndrome
Brief Title: A Safety Study of NNZ-2566 in Pediatric Rett Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuren Pharmaceuticals Limited (Industry)
Collaborators: rettsyndrome.org (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Neu-2566-RETT-002
Record Dates: First submitted 2016-02-21; First posted 2016-03-22 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Rett Syndrome
Keywords: Autism; Rett's syndrome; Rett disorder; Rett's disorder; Ataxia
MeSH Terms: conditions — Rett Syndrome; Autistic Disorder; Ataxia | interventions — trofinetide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NNZ-2566 (Experimental): Glycyl-L-2-Methylpropyl-L-Glutamic Acid
  Interventions: Drug: NNZ-2566
- Placebo (strawberry flavored solution) (Placebo Comparator): Strawberry flavored solution and Water for Injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNZ-2566 — Glycyl-L-2-Methylpropyl-L-Glutamic Acid (NNZ-2566) supplied as a lyophilized powder for reconstitution with strawberry flavored solution 0.5% v/v in Water for Injection.
  Other Names: trofinetide
  Arms: NNZ-2566
Drug: Placebo — Strawberry flavored solution and Water for Injection
  Other Names: Strawberry flavoring
  Arms: Placebo (strawberry flavored solution)

SUMMARY:
The purpose of this study is to determine whether NNZ-2566 is safe and well tolerated in the treatment of Rett syndrome in children and adolescents.

DETAILED DESCRIPTION:
Rett syndrome is a neurodevelopmental disorder primarily affecting females. The disorder is characterized by apparent normal development in early infancy (6-18 months), followed by a period of regression with onset of systemic and neurological signs. The CNS symptoms of Rett syndrome include learning disability, autism symptomatology and epilepsy and these can be severe and highly debilitating. Affected individuals also show signs of autonomic dysfunction, reflected in cardiovascular and respiratory abnormalities. There is no currently effective treatment for Rett syndrome.

This study will investigate the safety, tolerability and blood pharmacokinetics of treatment with oral administration of NNZ-2566 at 50 mg/kg, 100 mg/kg, 200 mg/kg BID, or placebo BID, in children and adolescent females with Rett syndrome. The study also will also investigate measures of efficacy and biomarkers during treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of classic/typical Rett syndrome with a documented mutation of the MeCP2 gene.
* Age 5 - 15 years.
* Weight at Screening and Baseline between 15.0 kg-100.0 kg (at least 15.0 kg and no greater than 100.0 kg).
* Each subject must be able to swallow the study medication provided as a liquid solution, or via gastrostomy tube.

Exclusion Criteria:

* Actively undergoing neurological regression
* Abnormal QT interval, prolongation or significant cardiovascular history.
* Current treatment with insulin.
* Anti-convulsants with liver enzyme inducing effects.
* Unstable seizure profile.
* Excluded concomitant medications.
* Current clinically significant (as determined by the investigator). cardiovascular, renal, hepatic, or respiratory disease.
* Gastrointestinal disease which may interfere with the absorption, distribution, metabolism or excretion of the study medication.
* History of, or current cerebrovascular disease or brain trauma.
* History of, or current clinically significant endocrine disorder, e.g. hypo- or hyperthyroidism, or diabetes mellitus.
* History of, or current, malignancy.
* Significant hearing and/or visual impairments that may affect ability to complete the test procedures.
* Allergy to strawberry.

Ages: 5 Years to 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
Adverse events | Through study completion, an average of 11 weeks
  Incidence of adverse events (AEs), including serious adverse events (SAEs), will be compared across the three NNZ-2566 doses and placebo. SAEs and AEs will be examined throughout the study.

SECONDARY OUTCOMES:
Motor Behaviour Assessment Scale (MBA) | Through study completion, an average of 11 weeks
Clinical Global Impression of Improvement (CGI-I) | Through study completion, an average of 11 weeks
Caregiver Top 3 Concerns via a Visual Analogue Scale (VAS) | Through study completion, an average of 11 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Glaze, MD, Principal Investigator — Baylor College of Medicine; Alan Percy, MD, Principal Investigator — University of Alabama at Birmingham; Timothy Feyma, MD, Principal Investigator — Gillette Children's Specialty Healthcare; Peter Heydemann, MD, Principal Investigator — Rush University Medical Center; Jeff Neul, MD, Principal Investigator — University of California, San Diego; Tim Benke, MD, Principal Investigator — Children's Hospital Colorado; Mary Jones, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland; Steve Skinner, MD, Principal Investigator — Greenwood Genetic Center; Mustafa Sahin, MD, Principal Investigator — Boston Children's Hospital; Sarika Peters, PhD, Principal Investigator — Vanderbilt University; Shannon Standridge, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Eric Marsh, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (12):
- United States (12):
  - University of Alabama, Birmingham, Alabama
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of California, San Diego, San Diego, California
  - Children's Hosptial Colorado, Aurora, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Greenwood Genetic Center, Greenwood, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Darwish M, Passarell J, Youakim JM, Bradley H, Bishop KM. Exposure-Response Efficacy Modeling to Support Trofinetide Dosing in Individuals with Rett Syndrome. Adv Ther. 2024 Apr;41(4):1462-1480. doi: 10.1007/s12325-024-02796-y. Epub 2024 Feb 16. PMID 38363467
- [Derived] Parent H, Ferranti A, Niswender C. Trofinetide: a pioneering treatment for Rett syndrome. Trends Pharmacol Sci. 2023 Oct;44(10):740-741. doi: 10.1016/j.tips.2023.06.008. Epub 2023 Jul 16. PMID 37460385